CLINICAL TRIAL: NCT01940757
Title: An Experimental Infection Study of Dermally-applied Infectious Necator Americanus Hookworm Larvae in Hookworm-naïve Adults
Brief Title: Experimental Infection of Hookworm-naïve Adults With Dermally-applied Infectious Necator Americanus Hookworm Larvae
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SVI-CH-01
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Hookworm Infection
Keywords: Necator americanus; Hookworm Infection; Experimental challenge infection
MeSH Terms: conditions — Hookworm Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (25 Necator americanus Hookworm Larvae) (Experimental): A dose of 25 Necator americanus Hookworm Larvae, administered via a sterile absorbent pad fixed with a transparent adhesive dressing for at least 1 hour.
  Interventions: Biological: Necator americanus Hookworm Larvae
- Cohort 2 (50 Necator americanus Hookworm Larvae) (Experimental): A dose of 50 Necator americanus Hookworm Larvae, administered via a sterile absorbent pad fixed with a transparent adhesive dressing for at least 1 hour.
  Interventions: Biological: Necator americanus Hookworm Larvae
- Cohort 3 (75 Necator americanus Hookworm Larvae) (Experimental): A dose of 75 Necator americanus Hookworm Larvae, administered via a sterile absorbent pad fixed with a transparent adhesive dressing for at least 1 hour.
  Interventions: Biological: Necator americanus Hookworm Larvae

INTERVENTIONS:
Biological: Necator americanus Hookworm Larvae — Infectious larvae of the human hookworm Necator americanus
  Other Names: Na-L3

SUMMARY:
An experimental hookworm infection model is being developed to provide early proof-of-concept that a hookworm vaccine targeting the blood-feeding pathway of adult hookworms is feasible and efficacious. The proposed model consists of vaccinating healthy, hookworm-naïve adults with a candidate hookworm vaccine, followed by challenging them with the investigational product, Necator americanus Larval Inoculum to assess the effect of vaccination on infection. The first proposed study will be a feasibility study that will consist of administering different doses of the Necator americanus Larval Inoculum to healthy adult volunteers to determine the optimal dose (i.e., number of infectious larvae) that is safe, well-tolerated and results in consistent infection.

DETAILED DESCRIPTION:
Open-label, dose-escalation clinical study in healthy, hookworm-naïve adults:

* Study site: George Washington Medical Faculty Associates, Washington, DC
* Number of participants: up to 35 in 3 cohorts

In Cohort 1, ten (10) volunteers will receive an inoculum of 25 infectious Necator americanus larvae. In Cohort 2, ten (10) volunteers will receive an inoculum of 50 infectious Necator americanus larvae. In the optional Cohort 3, fifteen (15) volunteers will receive an inoculum of 75 infectious Necator americanus larvae.

The cohorts will be enrolled in a staggered fashion with safety data assessed prior to larval dose escalation. Cohort 2 will be inoculated no earlier than 8 weeks after the last volunteer is inoculated in Cohort 1. The optional Cohort 3 will be inoculated no sooner than 8 weeks after the last volunteer is inoculated in Cohort 2. Cohort 3 will be enrolled only if the tolerability of the experimental infection of Cohort 2 is acceptable and does not result in significant adverse events.

Within each cohort, after Study Day 70, but before Study Day 77, up to 5 volunteers will undergo capsule endoscopy in order to visualize and count adult N. americanus hookworms residing in the intestine. Informed consent for capsule endoscopy will be obtained separately from the primary study, and agreement or refusal will not impact on a subject's eligibility to enroll or continue participation in the primary study.

Three months after larval administration, or at the time of study withdrawal, all participants will receive a 3-dose treatment of albendazole (400 mg per dose) for clearance of experimental infection.

* Larval inoculum schedule: Study Day 0 (single application)
* Route: applied to intact skin on the volar aspect of forearm
* Doses of N. americanus Larval Inoculum to be tested: 25, 50 and 75 infectious larvae (high dose optional)
* Study duration: 6 months per study participant; total duration of the study estimated at approximately 13 months
* Anthelmintic treatment: 3 months post larval inoculum, or at study withdrawal, 3-dose treatment with 400 mg albendazole

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 45 years, inclusive.
* Good general health as determined by means of the screening procedure.
* Available for the duration of the trial (6 months).
* Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

* Pregnancy as determined by a positive urine human choriogonadotropin (hCG) (if female).
* Participant unwilling to use reliable contraception methods while participating in the study (if female and not surgically sterile, abstinent or at least 2 years post-menopausal).
* Currently lactating and breast-feeding (if female).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
* Known or suspected immunodeficiency.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
* Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (hemoglobin <11.5 g/dl [females] or <12.5 g/dl [males]; absolute leukocyte count <3.6 or >10.7 x 103/mm3; absolute neutrophil count [ANC] <1.7 x 103/mm3; absolute lymphocyte count <0.7 x 103/mm3; or platelet count <140 x 103/mm3).
* History of iron deficiency anemia.
* History of hypoalbuminemia.
* Laboratory evidence of a coagulopathy (PTT or PT INR greater than 1.1-times the upper reference limit).
* Serum glucose (random) greater than 1.2-times the upper reference limit.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma as defined by the need for daily use of inhalers or emergency clinic visit or hospitalization within 6 months of the volunteer's expected Day 0 of the study.
* Positive ELISA for hepatitis B surface antigen (HBsAg).
* Positive confirmatory test for HIV infection.
* Positive confirmatory test for hepatitis C virus (HCV) infection.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of the volunteer's expected Day 0 of this study or planned use during the study.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to the volunteer's expected Day 0 of the study.
* Receipt of blood products within the past 6 months.
* Known allergy to amphotericin B or gentamicin.
* History of previous infection with hookworm or residence for more than 6 months in a hookworm-endemic area.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Study product-related adverse events | Up to 6 months after dosing
  Frequency of study product-related adverse events, graded by severity, for different doses of N. americanus Larval Inoculum.

SECONDARY OUTCOMES:
Fecal egg counts | Up to Study Day 101
  To determine the dose of N. americanus Larval Inoculum that generates the highest fecal egg counts, measured by fecal microscopy.
Number of adult hookworms in feces post-treatment | Study Days 87-101
  To compare the N. americanus Larval Inoculum dose received with the number of adult worms present in the gut, as determined by capsule endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: David J Diemert, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Diemert D, Campbell D, Brelsford J, Leasure C, Li G, Peng J, Zumer M, Younes N, Bottazzi ME, Mejia R, Pritchard DI, Hawdon JM, Bethony JM. Controlled Human Hookworm Infection: Accelerating Human Hookworm Vaccine Development. Open Forum Infect Dis. 2018 Apr 19;5(5):ofy083. doi: 10.1093/ofid/ofy083. eCollection 2018 May. PMID 29780848

DOCUMENTS (1):
  • Informed Consent Form (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT01940757/ICF_000.pdf